CLINICAL TRIAL: NCT05716347
Title: Safety and Immunogenicity of a Recombinant SARS-CoV-2 S-Trimer Vaccine (CHO Cell) as Booster Shots in Healthy Adults Aged 18-59 Years Who Have Completed Two Doses of Inactivated SARS-CoV-2 Vaccine
Brief Title: Clinical Trial of Safety and Immunogenicity of Recombinant SARS-CoV-2 S-Trimer Vaccine (CHO Cells) as Booster Vaccination in Populations Aged 18 to 59 Years
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Company strategy adjustment
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BS033VX-001
Record Dates: First submitted 2023-01-10; First posted 2023-02-08 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SARS-CoV-2 inactivated vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- the 5 μg recombinant SARS-CoV-2 S-Trimer vaccine booster group (Experimental)
  Interventions: Biological: the recombinant SARS-CoV-2 S-Trimer vaccine/inactivated SARS-CoV-2 vaccine
- the 10 μg recombinant SARS-CoV-2 S-Trimer vaccine booster group (Experimental)
  Interventions: Biological: the recombinant SARS-CoV-2 S-Trimer vaccine/inactivated SARS-CoV-2 vaccine
- the 30 μg recombinant SARS-CoV-2 S-Trimer vaccine booster group (Experimental)
  Interventions: Biological: the recombinant SARS-CoV-2 S-Trimer vaccine/inactivated SARS-CoV-2 vaccine
- ICV booster group (Active Comparator)
  Interventions: Biological: the recombinant SARS-CoV-2 S-Trimer vaccine/inactivated SARS-CoV-2 vaccine

INTERVENTIONS:
Biological: the recombinant SARS-CoV-2 S-Trimer vaccine/inactivated SARS-CoV-2 vaccine — one booster dose intramuscularly in the deltoid muscle of the upper arm.

SUMMARY:
Increased immune escape of emerging SARS-CoV-2 variants and waning neutralizing antibody levels over time indicate the importance of COVID-19 vaccine booster dose. Preclinical findings have shown that the recombinant SARS-CoV-2 S-Trimer vaccine exhibited favorable safety and immunogenicity. Herein, we conducted a randomized, open-label, positive control trial to assess the safety and immunogenicity of the booster shot in healthy subjects aged 18-59 years who have completed two-dose primary series of inactivated vaccine for 6-15 months. A total of 63 eligible participants were enrolled to receive the recombinant SARS-CoV-2 S-Trimer vaccine or inactivated vaccine, and only one participant in 30 μg recombinant SARS-CoV-2 S-Trimer vaccine cohort withdrew owing to personal work reasons on September 26, 2022. Subjects in each dose group (5 μg, 10 μg, 30 μg recombinant SARS-CoV-2 S-Trimer vaccine) was randomly assigned to receive the experimental vaccine or inactivated vaccine in a 2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were those who completed the two-dose primary series of ICV for 6-15 months
* Voluntarily consented to participate in this trial
* Agreed to take effective contraceptive measures (women of childbearing potential) from signing the informed consent form to 12 months after booster vaccination.

Exclusion Criteria:

* History of allergy to any vaccine or its excipients;
* Presence of severe, uncontrollable or hospitalized diseases;
* History of major surgery within 3 months prior to enrollment;
* History of Severe Acute Respiratory Syndrome (SARS), Middle East Respiratory Syndrome (MERS) or COVID-19;
* Congenital or acquired immunodeficiency or autoimmune disease;
* Any acute diseases or acute attacks of chronic diseases within 7 days prior to enrollment;
* Receipt of any COVID-19 prophylactic medication other than primary series of ICV;
* Long-term receipt (>14 consecutive days) of glucocorticoids or other immunosuppressive agents within the past 6 months;
* Receipt of biological agents, immunopotentiators or immunosuppressants within the past 6 months;
* Receipt of blood or blood-related products within 3 months prior to vaccination;
* Administration of antipyretics, painkillers or antiallergics within 24 hours prior to vaccination;
* Participating or planning to participate in other clinical trials during the study period;
* Pregnant or lactating females, women of childbearing age of pregnancy test positive;
* Presence of any underlying disease or condition which, in the opinion of the investigator, may place the subject at unacceptable risk, is unable to meet the requirements of the protocol, or interfere with the assessment of vaccine response.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | within 30 minutes after booster immunization
  All adverse events within 30 minutes of booster immunization
Incidence of Treatment-Emergent Adverse Events | within 7 days of booster immunization
  Solicited local/systemic AEs within 7 days of booster immunization
Incidence of Treatment-Emergent Adverse Events | within 28 days of booster immunization
  Unsolicited local/systemic AEs within 28 days of booster immunization
humoral immunogenicity | On Day 14 and Day 28 after booster immunization
  The Geometric Mean Titer (GMT) of neutralizing antibody against Delta, Omicron BA.2.2 and Omicron BA.5.2 after the booster immunization
humoral immunogenicity | On Day 14 and Day 28 after booster immunization
  The Geometric Mean Fold Rises (GMFR) of neutralizing antibody against Delta, Omicron BA.2.2 and Omicron BA.5.2 after the booster immunization
humoral immunogenicity | On Day 14 and Day 28 after booster immunization
  The seroconversion rate of neutralizing antibody against Delta, Omicron BA.2.2 and Omicron BA.5.2 after the booster immunization

SECONDARY OUTCOMES:
humoral immunogenicity | On 3rd month, 6th month after booster immunization
  The Geometric Mean Titer (GMT) of neutralizing antibody against Delta, Omicron BA.2.2 and Omicron BA.5.2 after the booster immunization
humoral immunogenicity | On 3rd month, 6th month after booster immunization
  The Geometric Mean Fold Rises (GMFR) of neutralizing antibody against Delta, Omicron BA.2.2 and Omicron BA.5.2 after the booster immunization
The safety outcomes were the counts and percentages of AEs, including SAEs and AESIs within 12 months, changes in laboratory safety parameters on the 3rd day following booster vaccination in comparison to baseline. | 12 months
  The safety outcomes were the counts and percentages of AEs, including severe adverse events (SAEs) and adverse of special interest (AESIs) within 12 months, changes in laboratory safety parameters on the 3rd day following booster vaccination in comparison to baseline.

OTHER OUTCOMES:
exploratory endpoints | on 0, 14 days, 3 months, 6 months after booster immunization
  Proportion of CD4+ cell subsets
exploratory endpoints | on 0, 14 days, 3 months, 6 months after booster immunization
  Proportion of CD8+ cell subsets
exploratory endpoints | on 0, 14 days, 3 months, 6 months after booster immunization
  Expression level of IFN-γ

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided